CLINICAL TRIAL: NCT04648020
Title: A Phase 2b/3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Comparing the Efficacy and Safety of Clonidine Mucoadhesive Buccal Tablet to Placebo to Prevent Chemoradiotherapy-induced Severe Oral Mucositis in Patients With Oropharyngeal Cancer
Brief Title: Clonidine HCl MBT vs. Placebo to Prevent Chemoradiotherapy-Induced Severe Oral Mucositis in Oropharyngeal Cancer.
Acronym: VOICE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim Analysis did not meet the pre-defined threshold for efficacy of a 15% absolute difference in SOM prevention between Validive and placebo.
Sponsor: Monopar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MNPR-301-001
Record Dates: First submitted 2020-11-19; First posted 2020-12-01 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Chemoradiotherapy-Induced Severe Oral Mucositis
Keywords: Mucositis; Oropharyngeal Cancer; Clonidine; Chemoradiotherapy; Severe Oral Mucositis; Monopar; Oral Mucositis; Head and Neck Cancer; Oral Cavity; Oropharynx; Mouth Sores
MeSH Terms: conditions — Mucositis; Oropharyngeal Neoplasms; Stomatitis; Head and Neck Neoplasms; Oral Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo Mucoadhesive Buccal Tablet given daily during chemoradiotherapy
  Interventions: Drug: Placebo Mucoadhesive Buccal Tablet
- Clonidine HCl Mucoadhesive Buccal Tablet (MBT) (Experimental): Clonidine HCl MBT given daily during chemoradiotherapy
  Interventions: Drug: Clonidine HCl Mucoadhesive Buccal Tablet

INTERVENTIONS:
Drug: Clonidine HCl Mucoadhesive Buccal Tablet — 100 μg of clonidine per tablet
  Other Names: Validive®
  Arms: Clonidine HCl Mucoadhesive Buccal Tablet (MBT)
Drug: Placebo Mucoadhesive Buccal Tablet — Placebo
  Arms: Placebo

SUMMARY:
This study is being performed to evaluate the effectiveness of a new drug, clonidine HCl MBT, to prevent the onset of severe oral mucositis (SOM) in patients with oropharyngeal cancer (OPC) who are being treated with chemoradiotherapy. OPC occurs on the back of the tongue or throat and is often treated by the use of chemoradiotherapy, where radiation is localized to these areas. Radiation to the OPC affected tissues causes the release of small proteins called cytokines that cause damage to the area surrounding the tumor including the oral cavity. This damage is characterized by the formation of mucositis which includes redness, pain and ulcers in the mouth and back of the throat. In addition, as more chemoradiation is administered to treat OPC, the inability to eat a solid diet (a Grade 3 mucositis) or to consume anything at all by mouth (a Grade 4 mucositis) occurs in many patients. Collectively, Grade 3 and Grade 4 mucositis is referred to as SOM. It is a frequent, debilitating side effect of chemoradiation in OPC that may cause patients to stop or interrupt their treatment, develop other side effects like the inability to swallow, or require the increased use of pain medications. OPC survivors who have successful treatment of their tumors often develop permanent swallowing, speaking and range of motion issues that may be linked back to the inability to eat and/or drink caused by SOM during their chemoradiotherapy treatment. Clonidine may inhibit the production of cytokines that cause SOM and clonidine HCl mucoadhesive buccal tablet (MBT) has been designed to deliver sustained high levels of clonidine in the oral cavity, potentially decreasing cytokine production and leading to a decrease in the incidence of SOM. Clonidine HCl MBT is a once per day treatment provided as a tablet that a patient may self-administer to the gums, where it sticks tightly to release clonidine over many hours. The primary objective of this Phase 2b/3 study is to evaluate whether clonidine HCl MBT is more effective than placebo MBT in decreasing the incidence of SOM.

DETAILED DESCRIPTION:
This is a sequential design Phase 2b/3 multicenter, randomized (1:1), double-blind, placebo-controlled, parallel group study to compare the efficacy and safety of clonidine HCl MBT to placebo MBT in the prevention of severe oral mucositis (SOM) in patients with oropharyngeal cancer (OPC) undergoing chemoradiotherapy (CRT). Best supportive care (BSC) will be allowed as per individual institutional practice with some exceptions as described in the inclusion and exclusion criteria. Eligible patients will be randomized to receive either clonidine MBT or placebo. Patients will be centrally randomized in a 1:1 ratio. The randomization will be stratified by p16 status (positive or negative). Randomized patients will be required to self-apply the study drug to the gum once a day in addition to BSC. The first application of MBT study drug will be performed on Day 1 of the CRT regimen. Each site will require the patient to follow the same local practice for BSC per Multinational Association of Supportive Care in Cancer/International Society of Oral Oncology (MASCC/ISOO) guidelines with some exceptions as described in the inclusion and exclusion criteria. Daily, self-administered MBT study drug will be continued once daily for the entire duration of CRT treatment; defined as from Day 1 of CRT until the last day of CRT (anticipated to be approximately 4-8 weeks depending on the patient's prescribed CRT plan). Patients will be recruited sequentially into either the Phase 2b or the Phase 3 part of the study. An interim analysis will be conducted when Phase 2b patients have either completed their CRT or discontinued from the study. The Data Monitoring Committee (DMC) will review the Phase 2b efficacy and safety data at the interim analysis and will make a recommendation on proceeding with the Phase 3 part of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male/Female patients of ≥ 18 years of age. Patients with histologically or pathologically confirmed squamous cell carcinoma of the oropharynx (including tonsils or the base of tongue) at one or several sites.
2. Patients treated with surgical resection of their primary tumor for localized or locally advanced disease T ≥ T0 and/or N ≥ N1 without distant metastasis (M0) (American Joint Committee on Cancer - AJCC 8th edition) and initiating adjuvant concurrent CRT within 8 weeks post-operatively. Unknown primary with node-positive disease confirmed to be Squamous Cell Carcinoma would be allowed or Patients who will be treated with definitive concurrent CRT for locally advanced disease T ≥ T0 and/or N ≥ N1 M0 (American Joint Committee on Cancer - AJCC 8th edition).
3. Patients eligible to receive a continuous course of external fractionated irradiation [conventional or intensity modulated radiation therapy (IMRT)] based on a daily dosing of 1.8 to 2.2 Gy/day 5 days/week in combination with cisplatin monotherapy either every 3 weeks (100 mg/m2) or weekly cisplatin (40 mg/m2). Alternative treatment regimens are allowed only if cisplatin is contraindicated. The decision on which cisplatin regimen to use in combination with IMRT and study drug/placebo will be at the discretion of the investigator.
4. Radiation plan must include delivery of a cumulative dose of 60-72 Gy. The oropharynx should receive at least 50 Gy.
5. Patients with adequate laboratory values defined as:

   1. Absolute neutrophil count ≥ 1.5 × 10^9/L
   2. Platelet count ≥ 75 × 10^9/L
   3. Hemoglobin ≥ 9 g/dL
   4. Creatinine blood level ≤ 1.5 × upper limit of the normal range (ULN)
   5. Total bilirubin ≤ 1.5 × ULN; patients with Gilbert's Syndrome can be included if hyperbilirubinemia ≤ 3 × ULN
   6. Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN
6. Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. A performance status of 2 is allowed only if due to a patient's malignancy.
7. Patients must provide written informed consent.
8. Human Papillomavirus (HPV) status documented by immunohistochemical detection of p16 expression in the tumor.
9. Negative serum pregnancy test for females of child-bearing potential at screening. A female is eligible to enter and participate in the study if the female is of non-child-bearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had a hysterectomy, a bilateral oophorectomy (ovariectomy), a bilateral tubal ligation, or is post-menopausal with a minimum of 1 year without menses.
10. Males with female partners of child-bearing potential and females of child-bearing potential must agree to use effective contraception starting prior to the first day of study drug treatment and continuing for 3 months after the last dose of study drug MBT.
11. Patients must be willing to complete questionnaires on a tablet, home computer, or paper form.

Exclusion Criteria:

1. Patients with no tumor or lesion in the oropharynx.
2. Prior induction chemotherapy for treatment of current malignancy.
3. Patients with planned accelerated IMRT.
4. Evidence of a concomitant other malignancy and/or any prior malignancy without complete remission in the last 2 years, except adequately treated basal or squamous cell carcinoma of the skin or in situ cervical cancer.
5. Patients with OM at baseline, any other oral ulceration or active oral infection (e.g., aphthous ulcers, orofacial herpes). Patients with post-operative pain of the mouth or throat are eligible.
6. Patients with known human immunodeficiency virus (HIV) seropositivity, known active Hepatitis B or C or known active tuberculosis.
7. Patients with systolic blood pressure (BP) < 100 mmHg and/or diastolic BP < 50 mmHg.
8. Patients with symptomatic cardiac dysrhythmia.
9. Patients with recent (less than 6 months) acute cardiovascular diseases (i.e., stroke, myocardial infarction).
10. Patients with any clinical condition, psychiatric condition, or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with study requirements and follow-up visits.
11. Patients currently being treated with sultopride, clonidine hydrochloride (eg, Catapres®), pentoxifylline or pilocarpine.
12. Patients intended to be treated specifically to prevent OM with any of the following:

    a. Bioadherent agents and mouthwashes: i. GelClair (consists of polyvinylpyrrolidone, hyaluronic acid, and glycyrrhetinic acid) ii. Sucralfate iii. Episil mouth spray iv. MuGard oral mucoadhesive v. Saforis (L-glutamine (topical)) b. Drug therapies and biologics: i. Amifostine (and similar free radical scavenger/antioxidant medications) ii. Palifermin (recombinant human keratinocyte growth factor-(KGF-1)) iii. Glutamine b. Interventional therapies i. Low level laser therapy (LLLT)
13. Patients who are unable to tolerate oral diet and/or are feeding tube dependent at baseline.
14. Patients receiving an approved or an investigational anti-cancer agent other than those specified in this study.
15. Patients with a known hypersensitivity to clonidine or any of the MBT excipients.
16. Women who are pregnant or breast-feeding.
17. Patients whose medical, psychological or surgical conditions are unstable and may affect the study completion and/or compliance and/or the ability to give informed consent.
18. Men and women of child-bearing age and their respective partners unwilling to use a highly effective contraception method during the study and for 3 months after the last administration of study drug.
19. Patient who has participated in another clinical trial with an investigational drug in the last 30 days prior to randomization in the present clinical study.
20. Subjects with orthostatic hypotension, defined by a decrease of systolic BP and/or diastolic BP above 20 mmHg when the patient stands up.
21. Conditions including but not limited to COVID-19 which would confound the assessment of the effects and/or safety of study medication in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-14 (Actual)

PRIMARY OUTCOMES:
To demonstrate the efficacy of HCl MBT to prevent SOM in OPC patients receiving CRT. | From the first CRT treatment through the end of the study treatment period, which is estimated to be 7 weeks.
  The occurrence of SOM (Yes/No), defined as any reporting of World Health Organization (WHO) Grade 3-4 OM, from the first day to the last day of CRT. The WHO mucositis grading scale will be used to assess the occurrence of SOM in this trial. The WHO grading scale grades OM from 0 to 4 according to severity of clinical observation and functional limitation, with Grade 4 = oral alimentation impossible, Grade 3 = Oral ulcers, liquid diet only, Grade 2 = Oral erythema, ulcers, solid diet tolerated, Grade 1 = Oral soreness, erythema, and Grade 0 = normal, no mucositis (no signs, no symptoms).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Up to 1 year after the first dose
  Evaluate the safety and tolerability of administering HCl MBT to OPC patients receiving CRT by assessing the number and severity of treatment-emergent adverse events (TEAE) and specifically those TEAEs of special interest. Adverse events are graded and tabulated using NCI CTCAE v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Holli Carlson, Study Director — Monopar Therapeutics Inc.
Locations (74):
- United States (48):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Orange Coast Memorial Medical Center, Fountain Valley, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Grand Valley Oncology, Grand Junction, Colorado
  - Christiana Care Health Services, Newark, Delaware
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Miami Cancer Institute, Miami, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - University Cancer & Blood Center, Athens, Georgia
  - IACT Health (Centricity Research), Columbus, Georgia
  - Decatur Memorial Hospital, Decatur, Illinois
  - Edward Elmhurst Health, Elmhurst, Illinois
  - NorthShore University Health Systems, Evanston, Illinois
  - AMITA Health, Hinsdale, Illinois
  - UnityPoint Health, Cedar Rapids, Iowa
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - East Jefferson General Hospital, Metairie, Louisiana
  - Louisiana State University Health - Shreveport, Shreveport, Louisiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Cox Medical Centers, Springfield, Missouri
  - Summit Health, Florham Park, New Jersey
  - New York Cancer and Blood Specialists, New York, New York
  - Northwell Health, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Novant Health Cancer Institute - Forsyth, Winston-Salem, North Carolina
  - Summa Health System, Akron, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Mercy Health, Youngstown, Ohio
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists, Tulsa, Oklahoma
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - AHN Cancer Institute - Allegheny General, Pittsburgh, Pennsylvania
  - Mary Hillman Radiation Oncology Center at UPMC Shadyside, Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Charleston Oncology, Charleston, South Carolina
  - Ballad Health, Johnson City, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Eastern Virginia Medical School, Norfolk, Virginia
  - PeaceHealth, Bellingham, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
  - HSHS St. Vincent Hospital Cancer Centers at HSHS St. Vincent Hospital, Green Bay, Wisconsin
- France (11):
  - Institut Andree Dutreix / Centre de Cancerologie Dunkerque, Coudekerque-Branche, Dunkerque
  - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire Morvan / Centre Hospitalier Universitaire de Brest, Brest
  - Centre hopitalier intercommunal de Créteil, Créteil
  - Centre Hospitalier de Dax-Côte d'Argent, Dax
  - Clinique François Chénieux, Limoges
  - Hôpital Saint Joseph, Marseille
  - Centre Hospitalier Universitaire La miletrie, Nice
  - Institut Jean Godinot, Reims
  - CHU de Saint Etienne, Saint-Priest-en-Jarez
  - Institut Gustave Roussy, Desmoulins, Villejuif
- Germany (3):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
  - Klinikum Kassel GmbH, Kassel
  - Caritas Klinikum Saarbrucken St. Theresia, Saarbrücken
- Ponce Medical School Foundation, Ponce, Puerto Rico
- Spain (11):
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Universitario Cruces de Bilbao, Barakaldo, Bizkaia
  - Hospital Meixoeiro, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia Hospitalet (Hospital Duran i Reynals), Barcelona
  - Hospital Universitario Quirónsalud Madrid, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Universitari Son Llàtzer, Palma de Mallorca
  - Hospital Complejo Universitario de Navarra, Pamplona
  - Hospital de Donostia, San Sebastián
  - Hospital Clínico Universitario Santiago de Compostela, Santiago de Compostela